CLINICAL TRIAL: NCT03755245
Title: PET/CT Study of Biodistribution and Performance of the [68Ga]Ga-DOTA-Siglec-9 in Patients With Rheumatoid Arthritis,Vasculitis or Pulmonary Sarcoidosis, and Radiation Dosimetry, Pharmacokinetics, Biodistribution, Safety and Tolerability in Healthy Men
Brief Title: Biodistribution, Dosimetry and Performance of [68Ga]Ga-DOTA-Siglec-9 in Healthy and Patients With Rheumatoid Arthritis, Vasculitis or Pulmonary Sarcoidosis
Acronym: SIGLEC
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Anne Roivainen, Professor, Turku University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: T282/2018
Record Dates: First submitted 2018-11-23; First posted 2018-11-27 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Healthy Subjects; Rheumatoid Arthritis; Vasculitis; Pulmonary Sarcoidosis
MeSH Terms: conditions — Arthritis, Rheumatoid; Vasculitis; Sarcoidosis, Pulmonary

STUDY DESIGN:
Intervention Model Description: Whole-body distribution, plasma pharmacokinetics, radiation dosimetry, safety, tolerability and performance of [68Ga]Ga-DOTA-Siglec-9
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [68Ga]Ga-DOTA-Siglec-9 (Other): Intravenous 140 MBq bolus injection of [68Ga]Ga-DOTA-Siglec-9 radiopharmaceutical
  Interventions: Other: [68Ga]Ga-DOTA-Siglec-9

INTERVENTIONS:
Other: [68Ga]Ga-DOTA-Siglec-9 — Vascular Adhesion Protein 1 (VAP-1) targeted radiopharmaceutical

SUMMARY:
This study evaluates safety, tolerability, biodistribution and performance of the [68Ga]Ga-DOTA-Siglec-9 following a single intravenous administration in patients with active rheumatoid arthritis, vasculitis or pulmonary sarcoidosis as well as radiation dosimetry, plasma pharmacokinetics, biodistribution, safety and tolerability of the tracer in healthy volunteers.

DETAILED DESCRIPTION:
Vascular adhesion protein 1 (VAP-1) is an inflammation inducible endothelial cell molecule mediating leukocyte trafficking from blood into the sites of inflammation. Although VAP-1 plays important role in early phases of inflammation, its luminal expression on the endothelium will remain constant if the inflammation continues, which suggest VAP-1 as a promising target for molecular imaging of inflammation. We have previously shown that sialic acid-binding immunoglobulin-like lectin 9 (Siglec-9) is a VAP-1 ligand, and the gallium-68 labeled 1,4,7,10-tetraazacyclododecane-N,N´,N´´,N´´´-tetraacetic acid conjugated peptide ([68Ga]Ga-DOTA-Siglec-9) containing residues 283-297 from Siglec-9 can be used for PET imaging of inflammation in various experimental models. This first-in-human study evaluates safety, tolerability, biodistribution and performance of [68Ga]Ga-DOTA-Siglec-9 after single intravenous injection in six healthy volunteers, and in ten patients with active rheumatoid arthritis (RA), five patients with vasculitis and five patients with pulmonary sarcoidosis.

ELIGIBILITY:
Inclusion Criteria:

* Healthy 18-70 year-old men
* Male or female 18-70 year-old patients with active rheumatoid arthritis, vasculitis or pulmonary sarcoidosis

Exclusion Criteria:

* In healthy: ongoing infection/inflammation proven by blood or other tests
* In patients with rheumatoid arthritis: no treatment with disease-modifying anti-rheumatic drugs or biologic agents, and no corticosteroids for 2 weeks prior the study
* In patients with vasculitis: no immunosuppressives, and glucocorticoid less than 60 mg for 2 weeks or NSAIDs for 1 day prior the study
* In patients with pulmonary sarcoidosis: no corticosteroids for 1 week or NSAIDs for day prior the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2018-11-23 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Whole-body distribution of [68Ga]Ga-DOTA-Siglec-9 | within a day
  Knowledge how intravenously injected [68Ga]Ga-DOTA-Siglec-9 is distributed in human body

SECONDARY OUTCOMES:
Radiation dosimetry of [68Ga]Ga-DOTA-Siglec-9 | within a week
  Absorbed ionisation radiation dose in critical organs due to single intravenous 140 megabecquerel injection of [68Ga]Ga-DOTA-Siglec-9

CONTACTS AND LOCATIONS:
Overall Officials: Anne Roivainen, Professor, Principal Investigator — Turku University Hospital, Turku PET Centre
Locations (1):
- Turku University Hospital, Turku PET Centre, Turku, Finland

REFERENCES:
- [Derived] Dadson P, Yla-Outinen H, Kalliokoski K, Tuokkola T, Malaspina S, Koivumaki M, Viitanen R, Rajala N, Silvoniemi M, Tolvanen T, Nuutila P, Jalkanen S, Saraste A, Saaresranta T, Taimen P, Roivainen A. Proof-of-concept PET imaging of pulmonary sarcoidosis using VAP-1-targeted radiotracer [68Ga]Ga-DOTA-Siglec-9. Respir Res. 2025 Dec 19. doi: 10.1186/s12931-025-03455-8. Online ahead of print. PMID 41420234